CLINICAL TRIAL: NCT00420589
Title: A Study to Assess the Efficacy and Tolerability of Taranabant in Maintaining Weight Loss Induced by Diet in Obese Patients Followed by a 1-Year Extension
Brief Title: A Weight Maintenance Study in Obese Patients (0364-012)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The overall profile does not support development for obesity
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0364-012; 2006_512
Record Dates: First submitted 2007-01-05; First posted 2007-01-11 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
Keywords: Weight loss; Weight regain; Weight maintenance
MeSH Terms: conditions — Obesity; Weight Loss | interventions — N-(3-(4-chlorophenyl)-2-(3-cyanophenyl)-1-methylpropyl)-2-methyl-2-((5-(trifluoromethyl)pyridin-2-yl)oxy)propanamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Placebo Comparator): Arm 1: MK0364 Pbo capsules once daily
  Interventions: Drug: Comparator: placebo
- 2 (Experimental): Arm 2: MK0364 0.5 mg capsule once daily
  Interventions: Drug: taranabant
- 3 (Experimental): Arm 3: MK0364 1 mg capsule once daily
  Interventions: Drug: taranabant
- 4 (Experimental): Arm 4: MK0364 2 mg capsule once daily
  Interventions: Drug: taranabant

INTERVENTIONS:
Drug: taranabant — taranabant 0.5 mg capsule, 1 mg capsule, 2 mg capsule once daily. Treatment for 52 weeks.
  Arms: 2; 3; 4
Drug: Comparator: placebo — Placebo capsules once daily. Treatment for 52 weeks
  Arms: 1

SUMMARY:
To compare the effects of taranabant versus placebo on weight regain and weight maintenance after low calorie diet-induced weight loss in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a body mass index (BMI) between 30 kg/m² and 43kg/m² and has maintained a stable weight (+/- 3kg) for at least 3 months prior to study start
* Patient is male or female >=18 and <= 65 years of age
* Patient understands the study procedures and alternative treatments available
* Patient is able to read, understand and complete study questionnaires

Exclusion Criteria:

* Patient has a history or presence of a major psychiatric disorder
* Patient has a recent history (within 6 months prior to signing the informed consent) diagnosis/episode/recurrence of stroke, TIA or neurological disorder
* Patient has a history of seizures or is at high risk of developing seizures
* Patient has systolic blood pressure >160mm Hg or diastolic blood pressure > 100 mm Hg
* Patient has diabetes mellitus as defined by medical history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2006-10; Primary Completion 2008-02 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Body weight at 52 weeks, safety and tolerability. | 52 weeks

SECONDARY OUTCOMES:
Body weight, biochemical markers, blood pressure, waist circumference and patient reported outcomes at 52 weeks. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Wadden TA, Fujioka K, Toubro S, Gantz I, Erondu NE, Chen M, Suryawanshi S, Carofano W, Johnson-Levonas AO, Shapiro DR, Kaufman KD, Heymsfield SB, Amatruda JM. A randomized trial of lifestyle modification and taranabant for maintaining weight loss achieved with a low-calorie diet. Obesity (Silver Spring). 2010 Dec;18(12):2301-10. doi: 10.1038/oby.2010.67. Epub 2010 Apr 8. PMID 20379151